CLINICAL TRIAL: NCT07305896
Title: Efficacy and Safety of Minocycline in the Treatment of Intracerebral Hemorrhage: a Multicenter, Randomized, Open-label, Blinded Endpoint Clinical Study
Brief Title: Efficacy and Safety of Minocycline in the Treatment of Intracerebral Hemorrhage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Enhance
Record Dates: First submitted 2025-12-14; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Minocycline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive an initial dose of 200 mg of minocycline hydrochloride capsules in addition to medical therapy after randomization, followed by 100 mg orally every 12 hours for 7 days, totaling 14 administrations.
  Interventions: Drug: Minocycline
- Control group (No Intervention): The control group will only receive medical therapy after randomization.

INTERVENTIONS:
Drug: Minocycline — The experimental group will receive an initial dose of 200 mg of minocycline hydrochloride capsules in addition to medical therapy after randomization, followed by 100 mg orally every 12 hours for 7 days, totaling 14 administrations.
  Arms: Experimental group

SUMMARY:
This study plans to enroll 1248 patients with supratentorial ICH within 24 hours of onset across multiple stroke centers. After randomization, the control group will only receive medical therapy. The experimental group, after randomization, will receive an initial dose of 200 mg of minocycline hydrochloride capsules in addition to medical ttherapy, followed by 100 mg orally every 12 hours for 7 days, resulting in a total of 14 administrations. Both groups will be followed for 180 days to evaluate the efficacy and safety of minocycline in the treatment of ICH.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, regardless of gender;
2. Supratentorial ICH confirmed by brain CT scan;
3. No disability in the community before ICH (premorbid mRS≤1);
4. Neurological deficits related to the hematoma, with NIHSS score ≥ 6 and single-limb motor item score ≥ 2;
5. GCS score ≥ 6;
6. Able to initiate the first dose of minocycline within 24 hours of onset;
7. Signed and dated informed consent.

Exclusion Criteria:

1. Definite evidence of secondary ICH, such as structural abnormality, brain aneurysm, brain tumor, use of thrombolytic drugs;
2. Allergy to tetracycline antibiotics;
3. Use of vitamin A derivatives or steroid therapy within the past 3 months;
4. Concomitant infection requiring antibiotic treatment at admission;
5. Planned surgical intervention;
6. Life expectancy of less than 6 months due to comorbid conditions;
7. Severe hepatic and renal dysfunction, or AST and/or ALT >3 times the upper limit of reference range, or serum creatinine >265 μmol/L (> 3 mg/dL);
8. Bleeding tendency, including heparin use within the past 48 hours (APTT ≥ 35 s), oral warfarin (INR > 2), platelet count < 100 × 10⁹/L, or hereditary hemorrhagic diseases;
9. Known pregnancy or breastfeeding;
10. Patients being enrolled or having been enrolled in another clinical trial within the 3 months prior to this clinical trial;
11. A high likelihood that the patient will not adhere to the study treatment and follow-up regimen;
12. Patients unsuitable for enrollment in the clinical trial according to the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1248 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with favorable functional outcomes, defined as mRS 0-2 at 180 days. | 180 days
  Modified Rankin Scale (mRS) ranged from 0 to 6, a low value represents a better outcome.

SECONDARY OUTCOMES:
The proportion of patients with an mRS score of 0-1 at 180 days. | 180 days
  Modified Rankin Scale (mRS) ranged from 0 to 6, a low value represents a better outcome.
The proportion of patients with favorable functional outcome (mRS score of 0-2) at 90 days. | 90 days
  Modified Rankin Scale (mRS) ranged from 0 to 6, a low value represents a better outcome.
The proportion of patients with an mRS score of 0-1 at 90 days. | 90 days
  Modified Rankin Scale (mRS) ranged from 0 to 6, a low value represents a better outcome.
The distribution of mRS scores at 90 days and 180 days. | 90 days and 180 days
  Modified Rankin Scale (mRS) ranged from 0 to 6, a low value represents a better outcome.
The NIHSS scores after 7 days of treatment. | 7 days
  The NIHSS is an ordinal hierarchical scale to evaluate the severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores indicating a more severe deficit.

OTHER OUTCOMES:
The incidence of any adverse events during the study period. | 180 days
  Adverse events.
The incidence of serious adverse events during the study period. | 180 days
  Serious adverse events.
The incidence of minocycline-related adverse events during the study period. | 180 days
  Minocycline-related adverse events.
Mortality during the study period. | 180 days
  Mortality.